CLINICAL TRIAL: NCT05293496
Title: A Phase 1/1b Dose Escalation and Cohort Expansion Study of MGC018 in Combination With Checkpoint Inhibitor in Participants With Advanced Solid Tumors
Brief Title: A Study of MGC018 in Combination With MGD019 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGC018-02
Record Dates: First submitted 2022-02-12; First posted 2022-03-24 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Castration-Resistant Prostatic Cancer; Malignant Melanoma; Pancreatic Ductal Carcinoma; Hepatocellular Cancer; Epithelial Ovarian Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Melanoma; Carcinoma, Pancreatic Ductal; Liver Neoplasms; Carcinoma, Ovarian Epithelial; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort -1 (Experimental): vobramitamab duocarmazine at dose level -1 and lorigerlimab intravenously (IV) every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine; Biological: lorigerlimab
- Cohort 1 (Experimental): vobramitamab duocarmazine at dose level 1 and lorigerlimab IV every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine; Biological: lorigerlimab
- Cohort 2 (Experimental): vobramitamab duocarmazine at dose level 1 and lorigerlimab IV every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine; Biological: lorigerlimab
- Cohort 3 (Experimental): vobramitamab duocarmazine at dose level 2 and lorigerlimab IV every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine; Biological: lorigerlimab
- Cohort 4 (Experimental): vobramitamab duocarmazine at dose level 3 and lorigerlimab IV every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine; Biological: lorigerlimab
- Cohort 5 (Experimental): vobramitamab duocarmazine at dose level 4 and lorigerlimab IV every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine; Biological: lorigerlimab
- Cohort Expansion (Experimental): maximum tolerated dose of vobramitamab duocarmazine and lorigerlimab IV every 4 weeks
  Interventions: Biological: vobramitamab duocarmazine; Biological: lorigerlimab

INTERVENTIONS:
Biological: vobramitamab duocarmazine — Vobramitamab duocarmazine is an antibody drug conjugate (ADC) targeted against B7-H3.
  Other Names: MGC018
Biological: lorigerlimab — Lorigerlimab is a bispecific DART® molecule that binds PD-1 and CTLA-4.
  Other Names: MGD019

SUMMARY:
Study CP-MGC018-02 is a study of vobramitamab duocarmazine (MGC018) in combination with lorigerlimab (MGD019). The study is designed to characterize safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics, and preliminary antitumor activity. Participants with relapsed or refractory, unresectable, locally advanced or metastatic solid tumors including, but not limited to, metastatic castration-resistant prostate cancer (mCRPC), melanoma, pancreatic cancer, hepatocellular carcinoma (HCC), ovarian cancer, and renal cell carcinoma (RCC) will be enrolled.

Vobramitamab duocarmazine and lorigerlimab are administered separately on Day 1 of every 4-week (28-day) cycle at the assigned dose for each cohort. Participants who do not meet criteria for study drug discontinuation may receive study drugs for up to 2 years.

Tumor assessments are performed every 8 weeks (± 7 days) for the initial 6 months on study drugs, then every 12 weeks (± 21 days) until progressive disease (PD).

Participants will be followed for safety throughout the study. .

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability to provide and document informed consent and willing and able to comply with all study procedures.
* Participants diagnosed with advanced solid tumors including but not limited to metastatic castration-resistant prostate cancer, melanoma, pancreatic cancer, hepatocellular carcinoma, ovarian cancer and renal cell carcinoma.
* Participants have received approved therapies according to their diagnosis.
* Participants must have an available tumor tissue sample. A fresh tumor biopsy may be performed if no archival sample is available.
* Eastern Cooperative Oncology Group performance status of less than or equal to 2.
* Life expectancy of at least 12 weeks.
* Evidence of measurable tumor for evaluation
* Acceptable end organ function according to laboratory results.
* Patients must agree to use highly-effective contraception during the study, and not donate sperm or ova.

Exclusion Criteria:

* Any underlying medical or psychiatric condition impairing participant's ability to receive, tolerate, or comply with the planned treatment or study procedures.
* Another malignancy that required treatment within the past 2 years. Participants who have had curative therapy for non-melanomatous skin cancer, localized prostate cancer (Gleason score < 6), or carcinoma in situ are eligible for the study.
* Active viral, bacterial, or fungal infection requiring systemic treatment within 1 week of initiation of study drug. Participants are eligible after SARS CoV 2-related symptoms have fully recovered for ≥ 72 hours.
* History of immunodeficiency. Participants with HIV are eligible if they have a CD4+ count ≥ 300/µL, undetectable viral load, and maintained on antiretroviral therapy for a minimum of 4 weeks.
* Prior autologous/allogeneic stem cell or tissue/solid organ transplant
* Prior treatment with MGD009, enoblituzumab, or other B7-H3 targeted agents for cancer.
* Clinically significant cardiovascular disease, lung compromise, venous insufficiency, or gastrointestinal disorders.
* Participants with greater than Grade 1 peripheral neuropathy.
* Participants who have a history of severe adverse events (AEs) from immune checkpoint inhibitors (anti-PD-1, anti-PD-L1, or CTLA-4 inhibitors). All other AEs from prior immune checkpoint inhibitors must be resolved to Grade 1 or less. Participants with any grade neurologic toxicity from prior immune checkpoint inhibitors are excluded.
* Pleural effusion or ascites. Trace pleural or peritoneal fluid is not exclusionary.
* History of Guillain-Barre syndrome, myasthenia gravis, or other autoimmune sensory or motor neuropathies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 2 years
Number of participants with serious adverse events (SAEs) | Up to 2 years
Number of participants with AEs leading to study treatment discontinuation | Up to 2 years

SECONDARY OUTCOMES:
Mean maximum observed concentration (Cmax) of vobramitamab duocarmazine | Throughout the study, up to 2 years
  Peak concentration of vobramitamab duocarmazine
Mean maximum observed concentration (Cmax) of lorigerlimab | Throughout the study, up to 2 years
  Peak concentration of lorigerlimab
Mean time to maximum concentration (Tmax) of vobramitamab duocarmazine | Throughout the study, up to 2 years
  Time at which peak concentration of vobramitamab duocarmazine is observed
Mean time to maximum concentration (Tmax) of lorigerlimab | Throughout the study, up to 2 years
  Time at which peak concentration of lorigerlimab is observed
Mean area under the concentration-time curve during the dosing interval (AUCtau) of vobramitamab duocarmazine | Throughout the study, up to 2 years
  Concentration of vobramitamab duocarmazine in the bloodstream during the 28-day dosing interval after dose administration
Mean area under the concentration-time curve during the dosing interval (AUCtau) of lorigerlimab | Throughout the study, up to 2 years
  Concentration of lorigerlimab in the bloodstream during the 28-day dosing interval after dose administration
Mean trough concentration of vobramitamab duocarmazine | Day 1 of each cycle (every 4 weeks) up to 2 years.
  Concentration of vobramitamab duocarmazine at the end of a dosing interval
Mean trough concentration of lorigerlimab | Throughout the study, up to 2 years
  Concentration of lorigerlimab at the end of a dosing interval
Number of participants who develop anti-drug antibodies (ADA) to vobramitamab duocarmazine | Throughout the study, up to 2 years
Number of participants who develop ADA to lorigerlimab | Throughout the study, up to 2 years
Objective response rate (ORR) | Assessed every 8 weeks for the first 6 months, then every 12 weeks for up to 2 years.
Median progression free survival (PFS) | Assessed every 8 weeks for the first 6 months, then every 12 weeks. Survival status is assessed approximately every 12 weeks after the last dose of study treatment until withdrawal of consent, lost to follow up, death, or end of the study, up to 2 years.
  PFS is defined as the time from the first dose date to the date of first documented PD or death from any cause, whichever occurs first.
Median duration of response (DoR) | Assessed every 8 weeks for the first 6 months, then every 12 weeks for up to 2 years.
  DoR is defined as the time from the date of initial response (CR or PR) to the date of first documented PD or death from any cause, whichever occurs first.
Median overall survival (OS) | Survival status is assessed approximately every 12 weeks after the last dose of study treatment until withdrawal of consent, lost to follow up, death, or end of the study, up to 2 years
  OS is defined as the time from the first dose date to the date of death from any cause.
Median radiographic PFS (rPFS) for mCRPC | Assessed every 8 weeks for the first 6 months, then every 12 weeks for up to 2 years.
  rPFS is defined as the time from the first dose of study drug to the first occurrence of radiographic PD of soft tissue lesions using RECIST v1.1, or appearance of ≥ 2 new bone lesions, or death from any cause
Prostate-specific antigen (PSA) response rate for mCRPC | PSA is assessed every 4 weeks, up to 2 years while on treatment, then every 12 weeks for up to an additional 2 years in follow-up.
  PSA response is defined as ≥ 50% decline from baseline in PSA with confirmation at least 3 weeks later.
Best PSA percent change from baseline for mCRPC | PSA is assessed every 4 weeks, up to 2 years while on treatment, then every 12 weeks for up to an additional 2 years in follow-up.
Median time to PSA progression for mCRPC | PSA is assessed every 4 weeks, up to 2 years while on treatment, then every 12 weeks for up to an additional 2 years in follow-up.
  PSA progression is defined as an increase that is ≥ 25% and ≥ 2 ng/mL the baseline or lowest value observed, and which confirmed by a second value at least 3 weeks later.
Median duration of PSA response for mCRPC | PSA is assessed every 4 weeks, up to 2 years while on treatment, then every 12 weeks for up to an additional 2 years in follow-up.
  DoR of PSA is defined as the time from the date of initial PSA response to the date of first documented PSA progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Casey, M.D., Study Director — MacroGenics
Locations (10):
- United States (10):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Florida Cancer Specialists and Research Institute, Sarasota, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Weill Cornell Medicine, New York, New York
  - Carolina BioOncology, Huntersville, North Carolina
  - Stephenson Cancer Center, The University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No